CLINICAL TRIAL: NCT01128751
Title: ELMAR - Elimination of Microemboli During Aortic Valve Replacement. A Randomized Controlled Trial
Brief Title: Elimination of Microemboli During Aortic Valve Replacement
Acronym: ELMAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Giessen (Other)
Collaborators: Else Kröner Fresenius Foundation (Other)
Responsible Party: PD Dr. Tibo Gerriets, Justus Liebig University, Department of Neurology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: P41/09// A67/09
Record Dates: First submitted 2010-05-18; First posted 2010-05-24 (Estimated); Last update posted 2010-05-24 (Estimated); Status verified 2010-05

CONDITIONS: Neurocognitive Outcome After Aortic Valve Replacement
Keywords: Cognition; Neuroprotection; Cardiopulmonary bypass; Aortic valve replacement; Micro-emboli
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Embol-X (Active Comparator): Patients in this arm receive intra-aortic filter designed to catch solid debris for neuroprotection during surgery.
  Interventions: Procedure: Embol-X intra-aortic emboli filter
- DBT dynamic bubble trap (Active Comparator): Patients in this arm receive a dynamic bubble trap to reduce gaseous micro-emboli from cardiopulmonary bypass for neuroprotection during surgery
  Interventions: Procedure: DBT dynamic bubble trap
- Control group (No Intervention): In comparison to arm 1 and 2, patients in this arm do not receive an additional intervention during surgery
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Embol-X intra-aortic emboli filter — Patients in this arm receive intra-aortic filter designed to catch solid debris for neuroprotection during surgery.
  Arms: Embol-X
Procedure: DBT dynamic bubble trap — Patients in this arm receive a dynamic bubble trap to reduce gaseous micro-emboli from cardiopulmonary bypass for neuroprotection during surgery
  Arms: DBT dynamic bubble trap
Procedure: Control group — In comparison to arm 1 and 2, patients in this arm do not receive an additional intervention during surgery
  Arms: Control group

SUMMARY:
In a randomized controlled trial patients undergoing aortic valve replacement are recruited into 3 groups. Patients receive either an intra-aortic filter (Embol-X), designed to reduce solid microemboli during mechanical surgical intervention, a dynamic bubble-trap (DBT), designed to reduce gaseous microemboli from cardiopulmonary bypass (CPB), or no additional device (control-group). Cognitive functioning is assessed 3 weeks to 1 day before and 3 months (+/- 1 week) after valve replacement. Furthermore, cerebral magnetic resonance imaging (MRI) is carried 2-6 days after surgery. Primary endpoint is the cognitive outcome of the filter groups compared to the controls. Secondary endpoint is the number of acute ischemic lesions after CABG.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Elective aortic valve replacement
* Informed consent
* German language

Exclusion Criteria:

* Neurological and psychiatric diseases that would conflict with neuropsychological testing (e.g. stroke, TBI, schizophrenia, etc.); further major surgeries on CPB planned for within 3 months after valve replacement
* Contraindication against MRI assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological assessment 1 | 3 weeks to 1 day before intervention
  Patients are assessed by an extensive neuropsychological test battery to test cognitive functions and psychological measures
Neuropsychological assessment 2 | 3 months (+/- 1 week) post intervention
  Patients are assessed by an extensive neuropsychological test battery to test cognitive functions and psychological measures

SECONDARY OUTCOMES:
MRI lesions detected after surgery | 2-6 days postoperative
  In MRI micro-embolic lesions are detected using diffusion weighted imaging (DWI)

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - University Clinic Giessen, 35392 Giessen, Hesse
  - Johann Wolfgang Goehte University Clinic, 60590 Frankfurt, Hesse
  - Kerckhoff Clinic, 61231 Bad Nauheim, Hesse